CLINICAL TRIAL: NCT02425293
Title: INCAS - Integrated Care of Asthma in Switzerland
Acronym: INCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hosptal, Baselland (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jörg Leuppi, Prof. Dr. med., Cantonal Hosptal, Baselland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 274/11
Record Dates: First submitted 2015-04-10; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients participating in a patient education seminar
  Interventions: Behavioral: asthma patient education
- Control (No Intervention): Patients not participating in a patient education seminar

INTERVENTIONS:
Behavioral: asthma patient education
  Arms: Intervention

SUMMARY:
The aim of this study was to investigate the effect of standardized patient education on asthma control. In collaboration with two health insurance companies, pharmacists and pneumologists, patients with asthma were recruited. They completed the "Asthma Control Test (ACT)" and the "Patient Assessment of Chronic Illness Care (PACIC 5A)" questionnaire to assess asthma control and patients' satisfaction with the health care service they received. Additionally, patients were offered the possibility to participate in a patient education seminar run by the Swiss lung leagues or the Swiss allergy centre (aha!). After one year, patients were asked to complete the questionnaires again. Comparisons of intraindividual changes and differences regarding ACT and PACIC 5A between patients with and without patient education were made.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical asthma diagnosis
* written informed consent

Exclusion Criteria:

* inadequate knowledge of the German language
* subjects with severe diseases with life expectancy under one year
* subjects with known Chronic Obstructive Pulmonary Disease (COPD)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 223 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Comparison of patient characteristics between the intervention and the control group | baseline
Comparison of asthma control between the intervention and the control group | baseline
  Asthma control is measured using the Asthma Control Test (ACT).
Comparison of patient satisfaction between the intervention and the control group | baseline
  Patient satisfaction is measured using the Patient Assessment of Chronic Illness Care (PACIC 5A) questionnaire.

SECONDARY OUTCOMES:
Comparison of asthma control at baseline and after one year in the intervention group. | baseline and follow up (after one year)
  Analysis of change in asthma control (using the Asthma Control Test (ACT)) in the intervention group from baseline to follow up (after one year).
Comparison of asthma control at baseline and after one year in the control group. | baseline and follow up (after one year)
  Analysis of change in asthma control (using the Asthma Control Test (ACT)) in the control group from baseline to follow up (after one year).
Comparison of patient satisfaction at baseline and after one year in the intervention group. | baseline and follow up (after one year)
  Analysis of change in patient satisfaction (using the PACIC 5A questionnaire) in the intervention group from baseline to follow up (after one year).
Comparison of patient satisfaction at baseline and after one year in the control group. | baseline and follow up (after one year)
  Analysis of change in patient satisfaction (using the PACIC 5A questionnaire) in the control group from baseline to follow up (after one year).